CLINICAL TRIAL: NCT01775488
Title: Safety and Initial Efficacy Study of the Vortx Rx for Treatment of Benign Prostatic Hyperplasia (Canada)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: HistoSonics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01.CP.0.2
Record Dates: First submitted 2013-01-21; First posted 2013-01-25 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Benign Prostatic Hyperplasia (BPH)
Keywords: Benign Prostatic Hyperplasia; BPH; LUTS; Vortx Rx; Histotripsy
MeSH Terms: conditions — Prostatic Hyperplasia

ARMS (1):
- Vortx Rx - Histotripsy BPH Device (Experimental): The Vortx Rx, is a portable ultrasound therapy device system that is intended for the treatment of BPH by using very intense, low duty-cycle ultrasound pulses to debulk prostatic tissue.
  Interventions: Device: Vortx Rx - Histotripsy BPH Device

INTERVENTIONS:
Device: Vortx Rx - Histotripsy BPH Device — Non-invasive histotripsy treatment / therapy to be delivered by surgeon using very low duty cycle ultrasound pulses from outside the patient's body. These pulses form a bubble cloud at the focal area within the prostate which mechanically breaks up the cellular structure of the soft tissue. During treatment, a surgeon is able to direct the bubble cloud throughout the targeted volume using controls located on the device console and using the real-time ultrasound for visualization feedback and control of the bubble cloud location.
  Other Names: HistoSonics Histotripsy BPH Device

SUMMARY:
The HistoSonics' Histotripsy BPH Device, the Vortx Rx, is a portable ultrasound therapy device. The purpose of this study is to assess and monitor the performance of the Vortx Rx for initial safety and efficacy for the treatment of Benign Prostatic Hyperplasia.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of BPH and eligible for endoscopic BPH surgery including Transurethral Resection of the Prostate [TURP], PVP, electrovaporization
2. Prostate volumes 30 - 80 gm based on transrectal ultrasound
3. Men ≥ 50 years of age
4. IPSS symptom score > 15 and IPSS bother score > 2
5. Baseline peak flow rate Qmax < 12 cc/s on two separate occasions with voided volume at least 150 cc

Exclusion Criteria:

1. History of prostate or bladder cancer, pelvic radiation, untreated bladder stones, urethral strictures/bladder neck contracture (BNC), renal insufficiency (i.e. creatinine > 1.4)
2. Neurogenic bladder, Parkinson's disease
3. Prior treatment for urinary incontinence
4. Micturition frequency AND urgency. Micturition frequency defined as > 8 micturitions per 24 hours as assessed by a thorough subject history including the question: "On average, how many times do you void during a 24 hour period? // < 4, 5-7, 8 or more." Urgency defined as an uncontrollable urge to void that occurs > 3 per 24 hours as assessed through the subject history/question: "On average, how many times a day do you have an uncontrollable urgency to void? // 0, 1-2, 3 or more?"
5. Intravesical prostate lobe protrusion > 1 cm on TRUS. Note: this is distinct from lateral lobes protruding up to the bladder such as an intravesical protrusion without median lobe
6. Active Urinary Tract Infection [UTI] (i.e. must have a screening urinalysis without signs of infection or a negative urine culture)
7. PVR > 250 at time of enrollment or catheter dependent bladder drainage
8. History of chronic prostatitis within the last 5 years
9. Not able to temporarily discontinue aspirin, Coumadin, Plavix and any other anticoagulant at least seven days prior to the time of treatment
10. History of known bleeding disorders (e.g. von Willebrand disease)
11. Prior BPH prostate procedures (e.g. Transurethral Microwave Therapy [TUMT], TUNA, water induced thermotherapy, TURP, PVP)
12. Men with confirmed or suspected malignancy of the prostate based on a digital rectal exam (DRE), prostate biopsy or PSA > 10 ng/mL. Men with free PSA < 25% and with PSA within an age and race-specific range may only be enrolled after a negative biopsy. If a biopsy is required, the subject shall have a six-week waiting period between the biopsy and histotripsy treatment, if he is deemed eligible to participate in the study.
13. Men interested in future fertility
14. Declines or unable to provide informed consent
15. Non-English-speaker
16. Life expectancy estimated to be less than one year
17. Unable or unwilling to complete all required questionnaires and follow-up assessments
18. In the opinion of the investigator, it is not in the subject's best interest to participate in the study.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-06; Primary Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | Up to 6 months
  * Record and report all adverse events.
  * Determine rate of occurrence of adverse events,serious adverse events and device-related adverse events as a measure of safety and as factors used to determine study success.

SECONDARY OUTCOMES:
Assess initial prostate histotripsy treatment efficacy | Up to six months
  1. Change in Lower Urinary Tract Symptoms [LUTS], International Prostate Symptom Score [IPSS], uroflow (Qmax), post-void residual (PVR). Each to be measured at 1, 3 and 6 months post-treatment
  2. Change in prostate parenchymal volume including TRUS and Prostate-Specific Antigen [PSA]. TRUS to be performed at end of treatment and at 6 months post-treatment. PSA to be tested at 6 months post-treatment.